CLINICAL TRIAL: NCT03389789
Title: Cortical Pain Processing in Full Term Infants, After Giving Different Non-pharmacological Analgesia
Brief Title: Newborn Cortical Response to Pain and Non Pharmacological Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC 50/11
Record Dates: First submitted 2017-12-27; First posted 2018-01-04 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Analgesia
Keywords: pain; infant; near-infrared spectroscopy; non pharmacological analgesia
MeSH Terms: conditions — Agnosia; Pain | interventions — Lactation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oral glucose solution + maternal holding (Experimental): Infants will receive 2 mL of oral glucose solution two minutes before the heel-prick and will be held in the mothers' lap (maternal relationship) throughout the painful procedure.
  Interventions: Other: Oral glucose solution + maternal holding
- Breastfeeding (Experimental): Infants will be breastfed two minutes before the heel-prick and throughout the painful procedure.
  Interventions: Other: Breastfeeding
- Oral glucose solution (Active Comparator): Infants will receive 2 mL of oral glucose solution given two minutes before the heel-prick on a changing table.
  Interventions: Other: Oral glucose solution
- Oral expressed breastmilk (Active Comparator): Infants will receive 2 mL of expressed breastmilk given two minutes before the heel-prick on a changing table.
  Interventions: Other: Oral expressed breastmilk

INTERVENTIONS:
Other: Oral glucose solution + maternal holding — Infant will receive both the oral glucose solution and the contact with the mother
  Arms: Oral glucose solution + maternal holding
Other: Breastfeeding — Infants will be breastfed
  Arms: Breastfeeding
Other: Oral glucose solution — Infant will receive only oral glucose solution without contact with the mother
  Arms: Oral glucose solution
Other: Oral expressed breastmilk — Infant will receive only oral expressed breast milk without contact with the mother
  Arms: Oral expressed breastmilk

SUMMARY:
Minor painful procedures are frequently performed on newborn infants and non-pharmacological analgesia is commonly used. As more than one analgesic method may be applied simultaneously in clinical practice, the relative contribution and efficacy of analgesic components still needs to be further elucidated. In the present study neonatal cortical brain response during four types of non-pharmacological analgesia (oral glucose, expressed breastmilk, maternal holding plus oral glucose, maternal holding plus breastfeeding) will be studied. The aim is to assess the differential effect of oral solutions (glucose, breastmilk), when given alone or in combination with maternal relationship (holding, breastfeeding). The study will test the hypothesis that the mother-infant relationship would improve the analgesic effect of oral solutions.

ELIGIBILITY:
Inclusion Criteria:

* Full term healthy infants, needing a heel-prick for metabolic screening;
* Informed consent obtained from parents.

Exclusion Criteria:

- Presence of sedation or analgesia (other than non pharmacological analgesia given during the experimental procedure)

Ages: 3 Days to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Cortical oxy-haemoglobin increase | During the procedure
  Multichannel near-infrared spectroscopy will be used to estimate cerebral cortex activation by measuring increase in cortical oxy-haemoglobin (HbO2)

SECONDARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS) | During the procedure
  The NIPS assesses 5 behavioral factors (facial expression, cry, arms, legs, and state of arousal) and one physiological factor (breathing patterns), each of which contains two items that are assigned scores of 0 or 1 (except for the crying factor, which comprises three items and is scored on a scale of 0 to 2). The scale yields a total score ranging from 0 to 7, where scores more than 3 are indicative of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Barbone, Prof, Study Chair — Institute for maternal and child health - IRCCS "Burlo Garofolo", Trieste, Italy; Stefano Bembich, MSC, Principal Investigator — Institute for maternal and child health - IRCCS "Burlo Garofolo", Trieste, Italy

REFERENCES:
- [Background] Bembich S, Cont G, Causin E, Paviotti G, Marzari P, Demarini S. Infant Analgesia With a Combination of Breast Milk, Glucose, or Maternal Holding. Pediatrics. 2018 Sep;142(3):e20173416. doi: 10.1542/peds.2017-3416. PMID 30166366